CLINICAL TRIAL: NCT06317922
Title: Evaluation of Dry Eye Disease's Signs in Patients Who Were Administered Intravitreal Injections
Brief Title: Evaluation of Dry Eye Disease's Signs in Patients Who Were Administered Intravitreal Anti-VEGF Injections
Acronym: DRYEYE-IVT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Francesco Bandello (Other)
Responsible Party: Sponsor-Investigator, Francesco Bandello, Full Professor and Chairman of Department of Ophthalmology, IRCCS Ospedale San Raffaele
Organization: IRCCS Ospedale San Raffaele (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DRYEYE-IVT Project
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Dry Eye Syndromes
Keywords: ocular surface discomfort
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: The participants will be randomized in two arms (treatment arm and control arm) in a ratio of 1:1.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: There are two teams:
  1. MASKED TEAM: Sub-investigators and study coordinators delegated to perform the following tasks:
     * dispensation to the patient the Investigational medical device (Thealoz Duo) or saline solution (Hydrabak containing Sodium Chloride 0,9 g, Sodium Dihydrogen Phosphate Dihydrate, Disodium Hydrogen Phosphate Dodecahydrate);
     * accountability of Investigational medical device and saline solution;
     * verify the compliance and therapeutic adherence of the patient;
     * discussion with the patient regarding the respect of the masked condition of the study;
  2. UNMASKED TEAMS:
     * informed consent process;
     * to perform the follow-up visit and assessments provided to test the ocular surface.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment arm (Experimental): Installation of artificial tears of Thealoz DUO (Investigational medical device containing trehalose 3 g and hyaluronic acid 0.15 g ), 10 ml.
  Dosage:1 drop x 4 times/day by 1 week before the Intravitreal injection until 3 months afterward.
  Interventions: Device: Thealoz Duo;
- control arm (Placebo Comparator): Installation of saline solution (Hydrabak containing Sodium Chloride 0,9 g, Sodium Dihydrogen Phosphate Dihydrate, Disodium Hydrogen Phosphate Dodecahydrate),10 ml.
  Dosage: 1 drop x 4 times/day by 1 week before the Intravitreal injection up to 3 months after it.
  Interventions: Device: sham (Hydrabak)

INTERVENTIONS:
Device: Thealoz Duo; — THEALOZ DUO is a solution containing trehalose (3%), sodium hyaluronate (0.15%), sodium chloride, trometamol, hydrochloric acid, and water for injections; Hydraback is a solution containing a sodium chloride 0.9 %, sodium dihydrogen phosphate dihydrate, sodium phosphate dodecahydrate, water for preparations for injection.
  Other Names: manufacturer: Laboratoires Théa; distributor: THEA Pharmaceuticals Ltd.
  Arms: treatment arm
Device: sham (Hydrabak) — Hydrabak is an ophthalmic solution containing: sodium chloride 0.9%, sodium dihydrogen phosphate dihydrate, sodium phosphate dodecahydrate, and water for injectable preparations
  Other Names: manufacturer: Laboratoires Théa; distributor: THEA Pharmaceuticals Ltd.
  Arms: control arm

SUMMARY:
The goal of this interventional, monocentric, prospective, single-masked, case-control study is to evaluate the efficacy of Thealoz Duo (artificial tear containing trehalose 3 g and hyaluronic acid 0.15 g) in comparison to a saline solution (Hydrabak containing Sodium Chloride 0,9 g, Sodium Dihydrogen Phosphate Dihydrate, Disodium Hydrogen Phosphate Dodecahydrate), to reduce the signs of ocular discomfort and ocular side effects in patients who have received Intravitreal injections.

The main questions it aims to answer are:

* can ocular instillation of Thealoz Duo solution, 1 week before intravitreal injection, in a fixed dose regimen, prevent ocular surface changes and dry-eye signs?
* can ocular instillation of Thealoz Duo solution, up 3 months after intravitreal injections, in a fixed dose regimen, reduce ocular surface changes, and dry-eye signs with improvement of quality of life and quality of vision?

Each participant will be randomized into each of two arms:

1. TREATMENT ARM: patients who will receive the instillation of Thealoz Duo, 10 ml, 1 drop, 4 times/day;
2. CONTROL ARM: patients who will receive the instillation of saline solution (Hydrabak), 10 ml, 1 drop, 4 times /day;

The decision of inclusion of a control group should minimize the risk of breaking the blinding condition by affecting the consistency and reliability of the outcome's achievement.

In any case, the instillation of saline solution should not alter the ocular surface.

ELIGIBILITY:
Inclusion Criteria:

* patient with retinal disease who required anti-VEGF therapy via intravitreal injections;
* patient who has already received at least 2 anti-VEGF therapy via intravitreal injections in the study eye during the last 6 months before the baseline;
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* patient with naive retinal disease who has already received < 2 anti-VEGF therapy via intravitreal injections in the study eye;
* subjects with autoimmune pathologies involving the ocular surface (e.g.Sjögren's syndrome), dry eye syndrome, eyelid disease that can induce changes in ocular surface (e.g. entropion, ectropion, lagophthalmos, trichiasis, ptosis), with any other systemic disease that may confound the interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-05-12 (Estimated); Study Completion 2025-05-12 (Estimated)

PRIMARY OUTCOMES:
Administration of Ocular Surface Disease Index (OSDI) to the patient | 3 months and 1 week
  The primary outcome is to evaluate the improvement of the dry-eye signs and changes in the ocular surface in patients who have received the intravitreal injections through the administration of Ocular Surface Disease Index (OSDI) at baseline, at month 1 and month 3 after the intravitreal injections.

SECONDARY OUTCOMES:
administration of Visual Analog Scale for Pain to the patient | 3 months and 1 week
  The Visual Analogue Scale measures pain intensity and consists of a 10cm line, with two endpoints representing 0 ('no pain') and 10 ('pain as bad as it could be').
evaluation of matrix metalloproteinase 9 gene expression | 3 months and 1 week
  The secondary outcome is to evaluate the improvements of ocular surface and signs related to dry eye disease, through:
  -evaluation of matrix metalloproteinase 9 gene expression.
TearLab Osmolarity | 3 months and 1 week
  The secondary outcome is to evaluate the improvements of ocular surface and signs related to dry eye disease, through:
  -TearLab Osmolarity.
Schirmer's test | 3 months and 1 week
  The secondary outcome is to evaluate the improvements of ocular surface and signs related to dry eye disease, through:
  -Schirmer's test.
tear film Break Up Time (tBUT) | 3 months and 1 week
  The secondary outcome is to evaluate the improvements of ocular surface and signs related to dry eye disease, through:
  -tear film Break Up Time (tBUT).
conjunctival hyperemia according to Efron grading scale | 3 months and 1 week
  The Efron grading scale describe the severity of contact lens complications (grade 0: normal; grade 1: trace; grade 2: mild; grade 3: moderate; grade 4: severe).
fluorescein staining | 3 months and 1 week
  The secondary outcome is to evaluate the improvements of ocular surface and signs related to dry eye disease, through:
  -fluorescein staining.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Bandello, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele _O.U. Ophthalmology, Milan, Italy

REFERENCES:
- [Result] Cejka C, Kubinova S, Cejkova J. Trehalose in ophthalmology. Histol Histopathol. 2019 Jun;34(6):611-618. doi: 10.14670/HH-18-082. Epub 2019 Jan 9. PMID 30623968
- [Result] Chiambaretta F, Doan S, Labetoulle M, Rocher N, Fekih LE, Messaoud R, Khairallah M, Baudouin C; HA-trehalose Study Group. A randomized, controlled study of the efficacy and safety of a new eyedrop formulation for moderate to severe dry eye syndrome. Eur J Ophthalmol. 2017 Jan 19;27(1):1-9. doi: 10.5301/ejo.5000836. Epub 2016 Jul 20. PMID 27445067
- [Result] Laude A, Lim JW, Srinagesh V, Tong L. The effect of intravitreal injections on dry eye, and proposed management strategies. Clin Ophthalmol. 2017 Aug 16;11:1491-1497. doi: 10.2147/OPTH.S136500. eCollection 2017. PMID 28860698
- [Result] Dohlman TH, Lertsuwanroj B, D'Amico DJ, Ciralsky JB, Kiss S. Evaluation of signs and symptoms of ocular surface disease after intravitreal injection. Acta Ophthalmol. 2019 Dec;97(8):e1154-e1156. doi: 10.1111/aos.14146. Epub 2019 Jun 25. No abstract available. PMID 31237739
- [Result] Saedon H, Nosek J, Phillips J, Narendran N, Yang YC. Ocular surface effects of repeated application of povidone iodine in patients receiving frequent intravitreal injections. Cutan Ocul Toxicol. 2017 Dec;36(4):343-346. doi: 10.1080/15569527.2017.1291665. Epub 2017 Feb 28. PMID 28166657